CLINICAL TRIAL: NCT06231121
Title: Short-term Results With Faricimab After Multiple Sequential Treatment Switches Due to Resistance With Both Aflibercept and Ranibizumab in Neovascular Age-related Macular Degeneration
Brief Title: Switching to Faricimab in Neovascular Age-related Macular Degeneration Resistant to Both Aflibercept and Ranibizumab
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Staff Specialist, Rigshospitalet, Denmark
Other Study IDs: MULTISW-VAB1SHOT
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients who received intravitreal faricimab injections between May and September, in 2023. and conform the inclusion/exclusion criteria.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — The Injections were performed according to local standard protocol, that included the use of 2-3 drops of topical tetracaine anesthesia, use of eye speculum, topical 5% povidone-iodine disinfection, a 30G-needle, injection site 3.5 mm posterior from the limbus marked by calipers in supertemporal or inferotemporal quadrants, a sterile cotton tip tamponade at the site of injection after removal of the needle, and no post-procedure antibiotics.
  Other Names: Vabysmo (6 mg, 0.05 ml)

SUMMARY:
The goal of this retrospective single-center chart review is to establish the response rate, efficacy and safety of a single dose of intravitreal faricimab injection in real-world patients with aflibercept- and ranibizumab-resistant neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion criteria

* Presence of neovascular age-related macular degeneration (AMD) in the study eye
* Previous treatment with minimum 6 consecutive, monthly aflibercept (Eylea®) injections in the study eye without optimal treatment response, defined as persisting intraretinal fluid or subretinal fluid or both on optical coherence tomography scans
* Subsequently, a sequential switch to ranibizumab (Lucentis®), with minimum 1 injection, also without optimal response
* Finally, a sequential treatment switch from ranibizumab to faricimab.

Exclusion criteria

* Neovascular conditions other than AMD (e.g., choroidal neovascularisation due to other causes) or co-existence of other retinal disease in the study eye
* Significant optical media opacities that would result in poor imaging quality on OCT scans in the study eye
* Intraocular surgery in the study eye 3 months before or within 1 month after the treatment switch

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular age-related macular degeneration (AMD)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients responding to the treatment switch | 4 weeks
  Defined as reduction or disappearance of the intra- or subretinal fluid at 4 weeks following a single injection of faricimab

SECONDARY OUTCOMES:
Differences in patient characteristics between individuals responding and not responding to faricimab | 4 weeks
Changes in central retinal thickness after the treatment switch | 4 weeks
  Measured on optical coherence tomography (OCT) scans
Changes in pigment epithelium detachment (PED) height after the treatment switch | 4 weeks
  Measured on optical coherence tomography (OCT) scans
Changes in best-corrected visual acuity after the treatment switch | 4 weeks

OTHER OUTCOMES:
Frequency of ocular and systemic adverse events | 4 weeks
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, MD, PhD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Miklos Schneider, Glostrup Municipality, Denmark